CLINICAL TRIAL: NCT03382171
Title: The Impact of FoodforCare at Home on Quality of Life of Cancer Patients Undergoing Chemotherapy.
Brief Title: The Impact of a Home Delivered Meal Service in Cancer Patients During Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-3044
Record Dates: First submitted 2017-11-23; First posted 2017-12-22 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2019-04

CONDITIONS: Cancer; Malnutrition
MeSH Terms: conditions — Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FoodforCare group (Experimental): The intervention group will receive meals from FoodforCare at Home. The FoodforCare at Home concept consists of five to six small protein and energy enriched meals that will be delivered twice a week. After an individual intake, the composition of the dishes will be tailored to the needs of the patient in terms of composition, diet, taste, flavor and portion size. Besides the meals, patients in the intervention group will also receive an information leaflet about the importance of protein during treatment and how to reach their protein requirements.
  Interventions: Other: FoodforCare at home
- Usual care group (No Intervention): The control group will continue their usual diet for 3 weeks and have no restrictions to their diet.

INTERVENTIONS:
Other: FoodforCare at home — Five small protein rich meals that will be delivered twice a week for 3 weeks.
  Arms: FoodforCare group

SUMMARY:
Cancer patients receiving treatment such as chemotherapy experience a variety of symptoms that interfere with their appetite and their ability to eat and enjoy meals. Therefore, adapting meals in a way that responds to these symptoms might be a good strategy to improve patient satisfaction, nutritional status and hence, quality of life. In this vein, the investigators hypothesize that meals from FoodforCare at Home will contribute to the quality of life of cancer patients undergoing chemotherapy when compared to usual care.

DETAILED DESCRIPTION:
Cancer patients receiving treatment such as chemotherapy experience a variety of symptoms that interfere with their appetite and their ability to eat and enjoy meals. Several studies suggest that nutritional intake increases when the patient is satisfied about the quality of the meals. Therefore, adapting meals in a way that responds to these symptoms might be a good strategy to improve patient satisfaction, nutritional status and hence, quality of life. In this vein, the investigators hypothesize that meals from FoodforCare at Home will contribute to the quality of life of cancer patients undergoing chemotherapy when compared to usual care. Also, the investigators expect that this strategy will have a positive effect on patient satisfaction, other nutrition-related issues, including nausea and vomiting, on nutritional intake per se and hence, on the nutritional status. Additional benefits might include reduced use of medication, especially anti-emetics.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* diagnosed with cancer
* receiving chemotherapy according to a minimum schedule of every 2 weeks
* living within a 40 km radius around the Radboud University Nijmegen Medical Centre
* written informed consent

Exclusion Criteria:

* renal insufficiency (MDRD-GFR (glomerular filtration rate) < 60ml/min and/or proteinuria)*
* dementia or any other condition which makes it impossible to fill out questionnaires correctly
* unable to understand or speak Dutch
* depending on artificial nutrition in the form of Oral Nutritional Supplements, tube feeding or total parenteral nutrition
* swallowing or passage problems

  * proteinuria is defined in case of a protein creatinine ratio > 0.5g/10mmol or an albuminuria > 300mg/day. This is checked by default before the start of chemotherapy by the treating physician to decide whether or not the patient is eligible for receiving chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Quality of life and overall health status | 3.5 months
  EORTC-Quality of Life-C30 questionnaire filled in before chemotherapy, two times during chemotherapy and after chemotherapy. This questionnaire consists of 30 questions and a total score ranging from 0-100 is calculated based on these questions. The higher the score, the higher the quality of life of the patient.

SECONDARY OUTCOMES:
Nutritional intake | 3.5 months
  2-day food diary filled in before chemotherapy, two times during chemotherapy and after chemotherapy.
Muscle strength | 3.5 months
  Hand grip strength (kg) performed before chemotherapy, two times during chemotherapy and once after chemotherapy.
Nutritional status | 3.5 months
  Patient Generated Subjective Global Assessment (PG-SGA) performed before chemotherapy, two times during chemotherapy and once after chemotherapy.
Functional score | 3.5 months
  Karnofsky scale performed before chemotherapy, two times during chemotherapy and once after chemotherapy. This status is based on 11 levels and ranges from 0, indicating death, to 100, indicating no complaints or evidence of disease.
Quality of life caregiver | 3.5 months
  Caregiver Reaction Assessment (CRA) filled in before chemotherapy, two times during chemotherapy and once after chemotherapy. This questionnaire consist of 24 items in five subscales. All items are statements with a 5-point Likert scale (completely disagree-completely agree). All subscale scores are the average of the item scores, ranging from 1 to 5. There is no total score.
Medication use | 3 weeks
  Diary filled in during 3 weeks between 2 cycles of chemotherapy
Symptoms | 3 weeks
  Symptom diary filled in during 3 weeks between 2 cycles of chemotherapy
Patient satisfaction | 1 day
  Questionnaire filled in after 3 weeks of receiving meals. This is a self-developed questionnaire which does not have a total score. Each question will be analyzed separately. Questions consist of grading from 0-10 (the higher, the better the outcome) or with a 5-point Likert scale (completely disagree-completely agree).
Functional status | 3.5 months
  Short Physical Performance Battery (SPPB) performed before chemotherapy, two times during chemotherapy and once after chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Manon van den Berg, PhD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coa KI, Epstein JB, Ettinger D, Jatoi A, McManus K, Platek ME, Price W, Stewart M, Teknos TN, Moskowitz B. The impact of cancer treatment on the diets and food preferences of patients receiving outpatient treatment. Nutr Cancer. 2015;67(2):339-53. doi: 10.1080/01635581.2015.990577. Epub 2015 Feb 9. PMID 25664980
- [Background] Teunissen SC, Wesker W, Kruitwagen C, de Haes HC, Voest EE, de Graeff A. Symptom prevalence in patients with incurable cancer: a systematic review. J Pain Symptom Manage. 2007 Jul;34(1):94-104. doi: 10.1016/j.jpainsymman.2006.10.015. Epub 2007 May 23. PMID 17509812
- [Background] Campbell AD, Godfryd A, Buys DR, Locher JL. Does Participation in Home-Delivered Meals Programs Improve Outcomes for Older Adults? Results of a Systematic Review. J Nutr Gerontol Geriatr. 2015;34(2):124-67. doi: 10.1080/21551197.2015.1038463. PMID 26106985
- [Background] Dashti HS, Mogensen KM. Recommending Small, Frequent Meals in the Clinical Care of Adults: A Review of the Evidence and Important Considerations. Nutr Clin Pract. 2017 Jun;32(3):365-377. doi: 10.1177/0884533616662995. Epub 2016 Sep 1. PMID 27589258
- [Background] Marin Caro MM, Laviano A, Pichard C. Nutritional intervention and quality of life in adult oncology patients. Clin Nutr. 2007 Jun;26(3):289-301. doi: 10.1016/j.clnu.2007.01.005. Epub 2007 Mar 21. PMID 17368656
- [Background] Leedo E, Gade J, Granov S, Mellemgaard A, Klausen TW, Rask K, Astrup A. The Effect of a Home Delivery Meal Service of Energy- and Protein-Rich Meals on Quality of Life in Malnourished Outpatients Suffering from Lung Cancer: A Randomized Controlled Trial. Nutr Cancer. 2017 Apr;69(3):444-453. doi: 10.1080/01635581.2017.1283421. Epub 2017 Feb 17. PMID 28287324
- [Derived] IJmker-Hemink V, Lize N, Beijer S, Raijmakers N, Wanten G, van den Berg M. Lessons learned from a randomized controlled trial on a home delivered meal service in advanced cancer patients undergoing chemotherapy: a pilot study. BMC Nutr. 2021 Feb 16;7(1):4. doi: 10.1186/s40795-021-00407-5. PMID 33588932

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT03382171/Prot_SAP_000.pdf